CLINICAL TRIAL: NCT03514511
Title: Randomised, Double-blind, Placebo-controlled, Single and Multiple Ascending Dose Trial to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of LEO 138559 in Healthy Subjects and Subjects With Moderate to Severe Atopic Dermatitis
Brief Title: Safety and Tolerability of LEO 138559 in Healthy Subjects and Subjects With Atopic Dermatitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: LP0145-1315
Record Dates: First submitted 2018-04-11; First posted 2018-05-02 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2021-03

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Cohort 1 in healthy subjects (Experimental): LEO 138559 (dose regiment 1) or LEO 138559 placebo
  Interventions: Drug: LEO 138559; Drug: LEO 138559 placebo
- Cohort 2 in healthy subjects (Experimental): LEO 138559 (dose regiment 2) or LEO 138559 placebo
  Interventions: Drug: LEO 138559; Drug: LEO 138559 placebo
- Cohort 3 in healthy subjects (Experimental): LEO 138559 (dose regiment 3) or LEO 138559 placebo
  Interventions: Drug: LEO 138559; Drug: LEO 138559 placebo
- Cohort 4 in healthy subjects (Experimental): LEO 138559 (dose regiment 4) or LEO 138559 placebo
  Interventions: Drug: LEO 138559; Drug: LEO 138559 placebo
- Cohort 5 in healthy subjects (Experimental): LEO 138559 (dose regiment 5) or LEO 138559 placebo
  Interventions: Drug: LEO 138559; Drug: LEO 138559 placebo
- Cohort 6 in healthy subjects (Experimental): LEO 138559 (dose regiment 6) or LEO 138559 placebo
  Interventions: Drug: LEO 138559; Drug: LEO 138559 placebo
- Cohort 7 in healthy subjects (Experimental): LEO 138559 (dose regiment 7) or LEO 138559 placebo
  Interventions: Drug: LEO 138559; Drug: LEO 138559 placebo
- Cohort 8 in subjects with atopic dermatitis (Experimental): LEO 138559 (dose regiment 8) or LEO 138559 placebo
  Interventions: Drug: LEO 138559; Drug: LEO 138559 placebo
- Cohort 9 in subjects with atopic dermatitis (Experimental): LEO 138559 (dose regiment 9) or LEO 138559 placebo
  Interventions: Drug: LEO 138559; Drug: LEO 138559 placebo

INTERVENTIONS:
Drug: LEO 138559 — LEO 138559 is a compound in development at LEO Pharma A/S
Drug: LEO 138559 placebo — LEO 138559 placebo

SUMMARY:
The primary objective of this trial is to investigate the safety and tolerability of LEO 138559 in healthy subjects and subjects with moderate to severe atopic dermatitis.

The secondary objective of this trial is to study the pharmacokinetics and pharmacodynamics following administration of LEO 138559 to healthy subjects and subjects with moderate to severe atopic dermatitis.

Healthy subjects will be exposed to 7 different dose regimens of LEO 138559 (one dose regimen per subject).

Subjects with moderate to severe atopic dermatitis will be exposed to 2 different dose regimens of LEO 138559 (one dose regimen per subject).

ELIGIBILITY:
Inclusion Criteria:

For healthy subjects and subjects with atopic dermatitis:

* Males and females without childbearing potential.
* Age between 18 and 55, inclusive.
* Body mass index between 18 and 32 kg/m2, inclusive.
* Healthy apart from atopic dermatitis for the subjects presenting the disease.

For subjects with atopic dermatitis only:

* History of atopic dermatitis for more than 6 months.
* Female subjects with childbearing potential and male subjects with female partners with childbearing potential using highly effective contraception from start of the trial and until a period after the last administered dose of trial drug.

Exclusion Criteria:

For healthy subjects and subjects with atopic dermatitis:

* Any significant disease detected prior to enrolment.
* Subjects who are still participating in a clinical trial or who have participated in a clinical trial within 3 months prior to enrolment or within 5 times of the half-life of the experimental therapy, whichever is longer.
* Skin diseases that may interfere with the diagnosis of atopic dermatitis or assessment of the treatment.
* Use of tanning beds or phototherapy within 6 weeks prior to enrolment.
* Subjects with atopic dermatitis requiring more than 3 bleach baths from 4 weeks prior to screening until end of trial.
* Blood pressure or pulse rate outside of the normal range.

For subjects with atopic dermatitis only:

* Initiation of treatment of atopic dermatitis with prescription emollients during the screening period.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2018-05-07 (Actual); Primary Completion 2021-03-02 (Actual); Study Completion 2021-03-02 (Actual)

PRIMARY OUTCOMES:
Safety of LEO 138559 - numbers of subjects with adverse events | Day 1 to Day 120
Safety of LEO 138559 - number of adverse events | Day 1 to Day 120
Tolerability of LEO 138559 - number of local site reactions | Day 1 to Day 120

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — LEO Pharma
Locations (3):
- United Kingdom (3):
  - Investigational site, Leeds
  - Investigational site, Liverpool
  - LEO Pharma investigational site, Manchester

IPD SHARING:
Plan to Share IPD: No